CLINICAL TRIAL: NCT01612156
Title: Use of 2% Lidocaine Gel Versus Water Based Lubrication: Is There a Difference in Pain During and After Multi-channel Urodynamics?
Brief Title: Lubricant Versus Lidocaine Gel for Pain Control During Urodynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Begum Ozel, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS- 11- 00573
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Pelvic Floor Disorders
Keywords: Urodynamic testing; pelvic floor examination; Lidocaine gel; Surgical lubricant; Pain; Embarrassment
MeSH Terms: conditions — Pelvic Floor Disorders; Pain | interventions — phenylmercury borate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2% lidocaine gel (Active Comparator): Subjects in this arm will have all urethral catheters and urethral cotton tipped swabs prepared with 2% lidocaine gel before use in the examination.
  Interventions: Drug: 2% lidocaine gel
- water based lubricant (Active Comparator): Subjects in this arm will have all urethral catheters and urethral cotton tipped swabs prepared wtih water based lubricant before use in the pelvic floor examination.
  Interventions: Drug: Water based lubricant

INTERVENTIONS:
Drug: 2% lidocaine gel — 2% lidocaine gel will be used to coat the urethral catheters and cotton tipped swab before use during the examination.
  Other Names: Lidocaine Hydrochloride Jelly USP, 2%
  Arms: 2% lidocaine gel
Drug: Water based lubricant — Water based lubricant will be applied to all urethral catheters and cotton tipped swabs before use in the pelvic floor examination.
  Other Names: Surgilube (Savage Laboratories)
  Arms: water based lubricant

SUMMARY:
The purpose of this study is to determine a difference in patient reported pain levels before, during, and after multichannel urodynamics in patients treated with 2% lidocaine gel or water based lubricant. We hypothesize that lidocaine gel will decrease pain levels when compared to lubricant gel.

DETAILED DESCRIPTION:
The evaluation of the incontinent patient usually includes in and out catheterization for post void residual urinary volume, a cotton tipped swab test, and urodynamic testing. All of these evaluations require manipulation of the urethra by either a catheter or a cotton tipped swab. To minimize discomfort, water based lubricant or 2% lidocaine gel is often used to ease passage of the device into the urethra. In 2008, Harmanli et al. performed a randomized control trial showing use of 2% lidocaine gel significantly decreased pain during the cotton tipped swab test and in and out catheterization. However, data looking at cystourethroscopy in women suggests that 2% lidocaine gel does little to relieve discomfort over lubricant alone. There are no studies looking at whether 2% lidocaine gel decreases the pain associated with multichannel urodynamic testing when compared to using lubricant alone. The purpose of this study is to determine a difference in patient reported pain levels before, during, and after multichannel urodynamics in patients treated with 2% lidocaine gel or water based lubricant. We hypothesize that lidocaine gel will decrease pain levels when compared to lubricant gel.

This study design is a prospective double blinded randomized controlled trial.

Participants will be randomized to the 2% lidocaine gel or the lubricant gel group after informed consent is obtained and immediately before undergoing multichannel urodynamics. Sequentially numbered sealed opaque envelopes containing the identity of the study arm will be used for randomization. The urogynecology clinic nurse will prepare the selected gel (either the 2% lidocaine gel or the water based lubricant) on the procedure field without any identification. Since the gels look identical, both the examiner and the patient will be blinded to their assigned arm. The participant will undergo the standard clinic exam in standardized order, which consists of perineal/vulvar sensation exam, measurement of post void residual, cotton tipped swab test, pelvic organ prolapse quantification measurements, pelvic exam with speculum, bi-manual exam, and multichannel urodynamic testing. The study gel will be applied to the red robinson catheter for in and out catheterization, the cotton tipped swab, and the bladder catheter for multichannel urodynamic study. The participant will be asked for their pain level at specific points (before the start of the exam, after placement of the bladder catheter, immediately after completion of the study, 30 minutes after completion of the study) using the Wong-Baker pain scale. At the conclusion of the procedure, the participant will be given a short survey to complete about their expectations of the procedure and their pain level. The practitioner/investigator will also be given a short survey to complete at the end of the examination to assess their idea of the patient's comfort level during the procedure. Data will be entered into a database for analysis using the independent samples t test, the Mann-Whitney U test, and the chi square test.

We will specifically be using Lidocaine Hydrochloride Jelly USP, 2% and Surgilube (Savage Laboratories). Surgilube is a water based lubricating gel used during gynecologic exams. It is available in 5g individually wrapped sterile packets. Lidocaine gel is also readily available for use in the gynecologic clinics, available in 5ml individually wrapped sterile packets. Both are clear, viscous, odorless, gels that are visually identical. Currently both are used in the standard urogynecologic exam, depending on operator preference.

All patients scheduled for urodynamic testing will be invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older
* Scheduled to undergo multichannel urodynamic study
* Able to give informed consent
* Able to read and write in English or Spanish

Exclusion Criteria:

* Any contraindication to multichannel urodynamic study
* Allergy to water based lubricant or lidocaine
* Any active pelvic or lower urinary tract infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Sun, M.D., Principal Investigator — University of Southern California
Locations (1):
- LAC USC Womens clinic, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2% Lidocaine Gel | Water Based Lubricant
Started | 42 | 48
Completed | 40 (Contraindication to urodynamics (urinary tract infection) diagnosed after randomization) | 48
Not Completed | 2 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2% Lidocaine Gel | Water Based Lubricant | Total
Number analyzed (Participants) | 40 | 48 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (9.1) | 50.2 (9.4) | 51.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 48 | 88
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Latina/Hispanic | 38 | 45 | 83
  African American | 2 | 2 | 4
  Non-Hispanic Caucasian | 0 | 1 | 1
Language [Number; unit: participants]
  English | 5 | 10 | 15
  Spanish | 35 | 38 | 73
Parity [Median (Full Range); unit: births] | 3 [0 to 6] | 3 [0 to 8] | 3 [0 to 8]
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 31.1 (4.5) | 30.1 (4.7) | 30.6 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Pain During the Pelvic Floor Examination
Description: Subjects will be asked to report their pain level using the Wong Baker pain scale at the beginning of the exam, after a cotton tipped swab test, after the urodynamic catheters are placed in the urethra, and then 30 minutes after the completion of the exam.
  The Wong Baker pain scale ranges from 0 (no pain) to 10 (worst pain possible).
Time Frame: 30 minutes after completion of exam
Measure: Mean (Standard Deviation); unit: units on Wong Baker pain scale
Arm/Group | 2% Lidocaine Gel | Water Based Lubricant
Number analyzed (Participants) | 40 | 48
units on Wong Baker pain scale
  Pain at baseline | 0.4 (1.0) | 0.9 (2.2)
  Pain after cotton tipped swab test | 1.3 (1.5) | 3.6 (3.2)
  Pain after placement of urodynamic catheters | 1.4 (1.9) | 3.9 (3.0)
  Pain 30 minutes after study completion | 0.7 (1.2) | 1.2 (2.0)

2. Secondary Outcome: Embarrassment With Pelvic Floor Examination
Description: The participants will be asked to report their level of embarrasment during the exam using a Likert scale from 1 (no embarrassment) to 5 (most embarrasment possible) at 30 minutes after completion of the exam.
Time Frame: 30 minutes
Measure: Median (Full Range); unit: On 5 point Likert scale
Arm/Group | 2% Lidocaine Gel | Water Based Lubricant
Number analyzed (Participants) | 40 | 48
On 5 point Likert scale | 2 [1 to 4] | 2 [1 to 5]

ADVERSE EVENTS:
Time Frame: Time frame for adverse event recording was 7 days.
Arm/Group | 2% Lidocaine Gel | Water Based Lubricant
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/48
Other Adverse Events (participants affected / at risk) | 0/40 | 0/48

LIMITATIONS AND CAVEATS:
Our patient population represented a predominantly Latina/Hispanic population, and our results might not be generalizable to other populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes